CLINICAL TRIAL: NCT01405261
Title: Investigation on Safety, Tolerability, and Pharmacokinetics of Single Doses of a Long-acting GLP-1 Analogue in Healthy Male Subjects
Brief Title: Trial Investigating the Safety of NNC 0113-0987 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN9926-3894; U1111-1119-1560 (Other: WHO); 2011-000297-57 (EudraCT Number)
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NNC 0113-0987 (gastro) (Experimental)
  Interventions: Drug: oral NNC 0113-0987; Drug: oral placebo
- NNC 0113-987 (coated) (Experimental)
  Interventions: Drug: oral NNC 0113-0987; Drug: oral placebo
- NNC 0113-987 (i.v) (Experimental)
  Interventions: Drug: I.v. NNC 0113-0987

INTERVENTIONS:
Drug: oral NNC 0113-0987 — Subjects will be randomised to receive a single dose of NNC 0113-0987 at escalating dose levels. Progression to next dose will be based on safety evaluation.
  Arms: NNC 0113-0987 (gastro)
Drug: oral NNC 0113-0987 — Subjects will be randomised to receive a single dose of NNC 0113-0987 at escalating dose levels. Progression to next dose will be based on safety evaluation.
  Arms: NNC 0113-987 (coated)
Drug: I.v. NNC 0113-0987 — Subjects will be administered a single i.v (into the vein) dose. The treatment with NNC 0113-0987 will be open-label, and will not be randomised.
  Arms: NNC 0113-987 (i.v)
Drug: oral placebo — Subjects will be randomised to receive a single dose of placebo.
  Arms: NNC 0113-0987 (gastro); NNC 0113-987 (coated)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate safety, tolerability and pharmacokinetics (the exposure of the trial drug in the body) of single doses of NNC 0113-0987 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with good general health as judged by the investigator, based on medical history, physical examination including 12-lead electrocardiogram (ECG), vital signs, and blood and urinary laboratory assessments at the screening visit
* Body Mass Index (BMI) of minimum 18.5 and below 30 kg/m^2

Exclusion Criteria:

* Male subjects who are sexually active and not surgically sterilised, who or whose partner are unwilling to use two different forms of effective contraception, one of which has to be a barrier method (e.g. condom with spermicidal foam/gel/film/cream) for the duration of the trial and for 3 months following the last dose of trial medication
* The receipt of any investigational product within 90 days (or 5 half-lives of investigational drug, whichever is greater) prior to this trial (screening), or is currently enrolled in any other clinical trial
* Subjects with a history of or presence of cancer, diabetes, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders that might have impact on the current trial, as judged by the investigator
* Subjects who are known to have hepatitis or who are carriers of the Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies, or have a positive result to the test for Human Immunodeficiency Virus (HIV) antibodies
* History of chronic or idiopathic acute pancreatitis or amylase or lipase values above 3x upper normal range (UNR)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Overview of Treatment Emergent Adverse Events (AEs) | Up to 25 days after trial product administration

SECONDARY OUTCOMES:
Frequency of hypoglycaemic episodes | From screening (day 1-21 before trial product administration) and until completion of the post treatment follow-up visit (day 12-25 after trial product administration)
AUC0-240h; area under the NNC 0113-0987 concentration-time curve | From time 0 to 240 hours after a single oral or intravenous (i.v.) dose
AUC, area under the curve | From time 0 to infinity after a single oral or i.v. dose
Cmax; maximum concentration of NNC 0113-0987 in plasma | After a single oral or i.v. dose
The time to maximum concentration (tmax) of NNC 0113-0987 in plasma | After a single oral dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Nottingham, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com